CLINICAL TRIAL: NCT02008292
Title: Acetylcholine, Tobacco Smoking, Genes and Nicotinic Receptors
Acronym: nic_physo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1210010989/2000021470; 2R01DA015577-05 (NIH); K23DA045957 (NIH); R01DA038832 (NIH)
Record Dates: First submitted 2013-12-02; First posted 2013-12-11 (Estimated); Results first posted 2023-02-06 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Smoking; Schizophrenia
Keywords: smoking; schizophrenia; acetylcholine
MeSH Terms: conditions — Smoking; Schizophrenia | interventions — Physostigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- physostigmine and amphetamine (Experimental): There is only one arm to the study. All subjects will receive physostigmine and amphetamine.
  Interventions: Drug: Physostigmine

INTERVENTIONS:
Drug: Physostigmine — All subjects will receive physostigmine to induce elevated ACh levels in the brain.
  Other Names: IV physostigmine

SUMMARY:
The purpose of the study is to measure the sensitivity of NCFHEB binding to changes in endogenous acetylcholine levels in healthy smoking and nonsmoking subjects, and in schizophrenic smoking and nonsmoking subjects. We hypothesize that physostigmine-induced elevated ACh levels will lead to a reduction in the availability of nicotinic receptors for the binding of the radioligand. We hypothesize there will be greater increase in ACh level (or greater reduction in radio tracer binding) in smoking as compared to nonsmoking subjects. We hypothesize there will be greater increase in ACh level (or greater reduction in radio tracer binding) in smoking as compared to nonsmoking subjects with schizophrenia, but the extent of this change will be different than in controls.

We are also measuring the sensitivity of PHNO binding to changes in dopamine levels in healthy smoking and nonsmoking subjects before and after amphetamine challenge.

DETAILED DESCRIPTION:
* Magnetic resonance image. Within approximately two weeks of the PET study, anatomical MRIs will be acquired at the Yale University MRI Center. Subjects will be taken through a ferromagnetic metal detector before entering the scan room. The purpose of the MRI scan is to direct the region of interest placement on the lower resolution PET images. The T1 weighted images will be acquired on a 3 Tesla Siemens Scanner. There will also be an additional resting state scan with subjects in the scanner, eyes open, fixating on a cross.
* Physostigmine challenge Physostigmine will be administered as follows. Glycopyrrolate, a cholinergic antagonist that does not have central side-effects, will be administered prior to physostigmine challenge to block physostigmine peripheral side-effects (e.g. nausea). Subjects will receive 200 mcg /ml x 1 ml of glycopyrrolate through an IV. Physostigmine administered i.v. has a short half life of 20 min with peak plasma levels 20-30 min post administration. The same dose of physostigmine will be administered as in the preliminary data: 1.5 mg/hr for 1 hr. Vital signs, including systolic and diastolic blood pressure, heart rate and respiration rate, will be monitored before physostigmine and then at 10, 20, 30, 60 min after the beginning of the infusion and then hourly until the end of the study day. Subjects will be questioned before, during, and after physostigmine challenge about potential adverse reactions typical to this medication (nausea, upset stomach, etc., as in Risks section). [If there is a significant and persistent drop in subjects' heart rate (>15% for at least 1 min), the IV physostigmine infusion will be stopped but the subject will continue to be monitored and will be discharged at the discretion of the study doctor. In emergency situation, PET center protocol will be followed accordingly (on file with HIC).
* Amphetamine challenge On PHNO PET days, subjects will have a baseline PHNO scan and then will receive amphetamine by mouth (0.5mg/kg). Approximately 2.5 hours after amphetamine administration, subjects will be scanned with PHNO again.
* Positron emission tomography PET scans may be performed on the High Resolution Research Tomograph (HRRT, 2-3 mm resolution) or another similar camera. Venous catheters will be used for i.v. administration of the radiotracer, venous blood sampling of AChE activity, and for the administration of glycopyrrolate and physostigmine. A radial artery catheter will be inserted by an experienced physician before the PET scan to draw arterial blood samples for metabolite analysis and for determination of the fraction of plasma radioactivity unbound to protein. At the beginning of scan, the subject's head will be immobilized and a transmission scan will be obtained for attenuation correction. PET scans will be acquired using bolus or bolus to infusion administration of up to 10 millicuries of NCFHEB or PHNO. Dynamic images of radioactivity concentration are reconstructed with corrections for attenuation, normalization, random events, scatter, and deadtime. Subject motion is corrected automatically on an event-by-event basis with the Vicra motion tracking system. Vital signs (blood pressure, pulse and respiration) are collected prior to and during each PET scan. Urine pregnancy test will be again administered on the PET scan day prior to the initiation of any imaging procedures. Smoking abstinence, when appropriate, will also be confirmed for smoking subjects prior to PET scanning.

PET scanning will then proceed as following for each aim:

Aim 1. Subjects will be asked to come to the PET center on two separate days to participate in one NCFHEB PET scan each time to assess test retest reproducibility of binding parameters measured with the radiotracer.

Aim 2. Subjects will participate in one PET scan day. Aim 3. Subjects from Aim 2 who are able to continue smoking abstinence will be asked to come back for another PET scan after about 6-8 weeks of smoking abstinence.

Aim 4. Baseline NCFHEB PET imaging will be conducted followed by administration of physostigmine. Preferably, this will be done on the same day. However, at times there is not enough radiotracer or subject is not able to tolerate a longer scan day. Therefore, some subjects may complete the study over two separate days (preferably within 1 month apart based on the availability of PET scanning times and subject's schedule).

Aim 5. Baseline NCFHEB PET imaging will be conducted followed by administration of physostigmine. Preferably, this will be done on the same day. However, at times when there is not enough radiotracer or when a subject is not able to tolerate a longer scan day. Therefore, some subjects may complete the study over two separate days (preferably within 1 month apart based on the availability of PET scanning times and subject's schedule).

Control subjects may participate in more than 1 aim. For example, nonsmoking subjects may complete Aim 1 and if chose, participate in Aim 4. Thus, subjects may participate in up to 4 PET scans for this protocol.

Aim 7. Subjects from Aim 4 will be asked to participate in 2 PHNO PET scans and amphetamine administration.

ELIGIBILITY:
Inclusion Criteria:

* who are able to read and write
* who are able to give voluntary written informed consent
* have no current uncontrolled medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology
* have no history of a neurological or psychiatric disorder (DSMIV Axis 1 and 2) other than schizophrenia in schizophrenia subgroup
* have not regularly used any prescription, herbal or illegal psychotropic medications (e.g. antidepressants, antipsychotics, anxiolytics, ecstasy) in the past 6 months (controls).
* Subjects with schizophrenia have not used any herbal or illegal substances in the past 6 months (medication inclusion listed below in Aim 5)
* drink less than <21 drinks/week for women and less than <35 drinks per week for men
* have not used marijuana in the past 30 days and have not met criteria for dependence in the past 2 years
* If female, not pregnant or breast feeding
* If female of childbearing age, must use an acceptable method of birth control, as determined by the principal investigator
* do not suffer from claustrophobia or any MR contradictions
* willing to donate blood for genetic studies
* willing to be followed up monthly after study participation via phone or email contact

Exclusion Criteria:

* Presence of acute or unstable medical or neurological illness. Subjects will be excluded from the study if they present with any history of serious medical or neurological illness or if they show signs of a major medical or neurological illness on examination or lab testing including history of seizures, head injury, brain tumor, heart, liver or kidney disease, eating disorder, diabetes.
* Presence of an Axis I diagnosis other than nicotine dependence and schizophrenia (for schizophrenia subgroup) in the past 2 years
* Regular use of any psychotropic drugs including anxiolytics and antidepressants and other over-the-counter medications and herbal products within the last year, and none within the last month for healthy controls.
* Regular use of antidepressants or psychotropic over-the-counter medications and herbal products within the last year
* For subjects with Schizophrenia, use of SSRI's (Paxil, Prozac Zoloft, Lexapro and Celexa) and use of tricyclic anti-depressants, except for a minimal dose used to treat anything other than depression, per the Investigator's discretion.
* Pregnancy/Breast feeding
* Subjects with a pacemaker or other ferromagnetic material in body.
* Subjects with a sitting pulse rate >100 bpm will be excluded
* Subjects with hypertension defined as sitting systolic blood pressure of >160 mmHg and/or sitting diastolic blood pressure of >100 mmHg will be excluded. Those individuals with hypertension that is well controlled by medication (e.g., within the above mentioned range) are not excluded
* Specifically, we will exclude subjects who have any active clinically significant deviation from the normal range in their electrocardiogram (EKG). However, subjects who have abnormalities in their EKG but the condition has been present for a while and the study cardiologist has evaluated and feels comfortable with the condition, would not be excluded on the basis of their cardiac condition. Examples of conditions that may meet these criteria (e.g., condition has been present for a while) include but are not limited to T-wave abnormalities, atrial fibrillation, prolonged PR interval, and right bundle branch block.
* Subjects with an allergy to salicylates
* Subjects with history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year.
* Subjects with current, past or anticipated exposure to radiation in the work place
* Blood donation within eight weeks of the start of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cosgrove, PhD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Yale Magnetic Resonance Research Center, New Haven, Connecticut
  - Yale PET Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy controls and healthy smokers will be recruited from the community through advertisements as approved by the Yale University Human Investigations Committee (HIC). Interested individuals contacting the clinic by phone in response to advertisements are told that the information they give over the phone is written down and discussed by the research team.
Groups:
- Healthy Controls for 1210010989; Healthy Smoker Controls for 1210010989: men and women aged 18-60 years who are able to read and write who are able to give voluntary written informed consent have no current uncontrolled medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology have no history of a neurological or psychiatric disorder (DSMIV Axis 1 and 2) other than schizophrenia in schizophrenia subgroup have not regularly used any prescription, herbal or illegal psychotropic medications (e.g.
  antidepressants, antipsychotics, anxiolytics, ecstasy) in the past 6 months (controls) that in the PI's determination puts the subject at increased risk or interferes with the study outcome. Subjects with schizophrenia have not used any herbal or illegal substances in the past 6 months (medication inclusion listed below in Aim 5) drink less than <21 drinks/week for women and less than <35 drinks per week for men have not used marijuana in the past 30 days and have not met criteria for dependence in the past 2 years If female, not pregnant or breast feeding If female of childbearing age, must use an acceptable method of birth control, as determined by the principal investigator do not suffer from claustrophobia or any MR contradictions willing to donate blood for genetic studies willing to be followed up monthly after study participation via phone or email contact
Period: Overall Study
Arm/Group | Healthy Controls for 1210010989 | Healthy Smoker Controls for 1210010989
Started | 43 (Total expected Healthy Control 1210010989 = 50 participants) | 37 (Total expected Smoking Healthy Control 1210010989 = 50 participants)
Completed | 43 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls for 1210010989 | Healthy Smoker Controls for 1210010989 | Total
Number analyzed (Participants) | 43 | 37 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 37 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 28 | 28 | 56
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 1 | 4
  African American | 14 | 13 | 27
  Caucasian | 15 | 17 | 32
  Hispanic | 10 | 4 | 14
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 43 | 37 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change in Acetylcholine (ACh) Levels After Physostigmine Administration as Confirmed by PET Images.
Description: PET images will be obtained in healthy controls and smoker subjects after physostigmine administration. Change in ACh levels will be determined by change in binding potential of Norchloro-fluoro-homoepibatidine (NCFHEB)
Time Frame: first 150 minute scan at baseline, second 150 minute scan start 10 minutes post physostigmine administration
Population: 66 of 80 participants were analyzed in primary study as 14 had signed consent but did not fully complete aim (i.e. Medical DQ by MD prior to drug administration or Relapse in smoking cessation by participant or medical aline failure, participant unable reschedule. For primary measure we only included participants that voluntarily completed both primary measures successfully.
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- ACH Levels in Healthy Controls After Physostigmine Administration: Physostigmine: Healthy Controls will receive physostigmine to induce elevated ACh levels in the brain.
- ACH Levels in Smokers After Physostigmine Administration: Physostigmine: Smokers will receive physostigmine to induce elevated ACh levels in the brain.
Arm/Group | ACH Levels in Healthy Controls After Physostigmine Administration | ACH Levels in Smokers After Physostigmine Administration
Number analyzed (Participants) | 34 | 32
percentage of change | 5.9 (6.5) | 4.3 (8.4)

2. Primary Outcome: Change in Dopamine (DA) Levels After Amphetamine Administration as Confirmed by PET Images.
Description: PET images will be obtained in all subjects after amphetamine administration. Change in DA levels will be determined by change in binding potential of PHNO, a selective dopamine D2 receptor agonist.
Time Frame: first 120 min scan at baseline, second 120 scan 2.5 hours after amphetamine administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Healthy Controls After Dextroamphetamine; Healthy Smoker After Dextroamphetamine: Dextroamphetamine: Healthy Controls will receive dextroamphetamine to elevated elevated DA levels in the brain.
Arm/Group | Healthy Controls After Dextroamphetamine | Healthy Smoker After Dextroamphetamine
Number analyzed (Participants) | 34 | 32
percentage of change | 26.5 (6.5) | 19.6 (10)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during study and up to 72 hours after PET imaging. Subjects were given research assistant and MD immediate contacts following scan in case of adverse event occurring after discharged. All subjects vitals had returned within 10% to original baseline vitals and were cleared by MD for discharge.
Description: The investigator will report the following types of adverse events to the IRB: a) serious AND unanticipated AND possibly, probably or definitely related events; b) anticipated adverse events occurring with a greater frequency than expected; and c) other unanticipated problems involving risks to subjects or others. These adverse events or unanticipated problems involving risks to subjects or others will be reported to the IRB within 48 hours of it becoming known to the investigator.
Arm/Group | Healthy Controls for 1210010989 | Healthy Smoker Controls for 1210010989
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/37
Other Adverse Events (participants affected / at risk) | 0/43 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT02008292/Prot_SAP_000.pdf